CLINICAL TRIAL: NCT00563277
Title: Surgical Treatment of Concurrent Cataract and Primary Pterygium: A Randomized Control Trial
Brief Title: Surgical Treatment of Concurrent Cataract and Primary Pterygium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2004.274-T; HARECCTR0500012
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Pterygium; Cataract; Lenses, Intraocular
Keywords: Pterygium; Cataract; Intraocular lens power calculation accuracy
MeSH Terms: conditions — Pterygium; Cataract

INTERVENTIONS:
Procedure: combined pterygium and cataract operation
Procedure: pterygium excision followed by cataract operation

SUMMARY:
Pterygium is known to induce with-the-rule astigmatism. The corneal curvature along the long axis of the pterygium body is flattened. The excision of pterygium will result in steepening of the cornea and reduction of astigmatism. Therefore, the effect of pterygium excision on intraocular lens (IOL) power calculation has been examined in our previous study. The study confirmed that pterygium can cause alteration of IOL power.

The determination of IOL power for cataract surgery is usually calculated from IOL formula called SRK II formula. IOL power = A - (2.5 x AL)-(0.9 x K). Variable A denotes the A-constant of the intraocular lens which is dependent on the IOL material and refractive index. Other variables for input include axial length (AL) and keratometry (K). A larger K reading will result in a lower estimated IOL power and vice versa. Previous studies have documented simultaneous cataract and pterygium operation resulted in reasonable visual outcome without adjustment of IOL power.

With the presence of a pterygium, the cornea is flattened and lead to a reduction of K value and over-estimation of calculated IOL power. This randomized controlled trial is designed to compare the refractive outcomes of sequential and simultaneous pterygium and cataract operation.

Pterygium excision should be done with various adjuvant therapies to minimize recurrence. Our previous studies reliably demonstrated limbal conjunctival graft and mitomycin C were effective methods to achieve low pterygium recurrence. We use limbal conjunctival autograft as the adjuvant therapy in the current study because this method is safer to be performed either alone or in combination with phacoemulsification. We avoid using mitomycin C as the adjuvant therapy in order to minimize the possibility of intraocular toxicity due to seepage.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Primary pterygium > 2mm across corneal limbus [Measurement made from the imaginary line of surgical limbus to the most advance edge of the visible pterygium tissue] Concurrent visually significant cataract ( BCVA < 20/70 )
* Informed consent for both pterygium and cataract surgery

Exclusion Criteria:

* Temporal pterygium
* Double headed pterygium
* Previous ocular surgery in which conjunctival-limbal graft is not feasible
* Pterygium covering visual axis that preclude keratometric assessment
* History of scleritis or autoimmune diseases

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2004-10; Study Completion 2006-12 (Estimated)

PRIMARY OUTCOMES:
final refraction deviation from target | 1 and 3 months post cataract operation

SECONDARY OUTCOMES:
change of IOL power from pre-pterygium estimated power | 1 and 3 months post pterygium excision

CONTACTS AND LOCATIONS:
Overall Officials: Lulu Cheng, Dr, Principal Investigator — Department of DOVS, Prince of Wales Hospital/ The Chinese University of Hong Kong
Locations (3):
- China (3):
  - Alice Ho Miu Ling Nethersole Hospital, Hong Kong
  - Hong Kong Eye Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong